CLINICAL TRIAL: NCT04870918
Title: Self-care Intervention for Reducing Rehospitalization for Heart Failure: a Randomized Clinical Trial (SIHF)
Acronym: (SIHF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Universidade de Caxias do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UP 5630/19
Record Dates: First submitted 2020-11-17; First posted 2021-05-04 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure
Keywords: heart failure; self-care; rehospitalisation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: One group will have self-care guidelines and the other will not. Medical appointments will be the same for both groups.
Who Masked: Outcomes Assessor
Masking Description: There will be blinding to assess outcomes, that is, review of medical records and phone calls in order to have knowledge about rehospitalization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self-care intervention (Experimental): First, health education will be carried out by the nurse. The consultations will be individual, weekly (Wednesdays), the others, therefore, will be biweekly, extending to the 30/30 days the following, individually in order to observe the difficulties and doubts of each patient. Counting the meetings in a total of 12 in the first 6 months.
  Interventions: Behavioral: self-care intervention
- usual care (No Intervention): The control group will go through medical consultations as instructed by the doctor and will not receive intervention for health education by the nurse.

INTERVENTIONS:
Behavioral: self-care intervention — Health education will be carried out by the nurse.
  Arms: self-care intervention

SUMMARY:
Introduction: Heart failure (HF) is considered an epidemic with high morbidity and mortality that imposes limitations on affected individuals, decreases the quality of life, restricts social life and makes it difficult to carry out daily activities including work. Almost 50% of diagnosed patients are readmitted in less than 90 days after discharge. Therefore, rehospitalization is considered as a predictive cause of the increased risk of intrahospital death in patients hospitalized with HF due to underlying disease. Related to chronic diseases, self-care is essential in maintaining physical and psychological well-being because it corroborates the success of the treatment. The patient's observational and resolving capacity is necessary in view of the appearance of signs and symptoms that would be postponed or alienated and would end up in hospital. Objective: To verify whether an intervention focused on self-care reduces the number of readmissions, improves quality of life and provides greater post-traumatic growth in patients with HF. Method: Randomized clinical trial, parallel by intention to treat, with blinding for evaluation of outcomes. Adult patients who were admitted to a Hospital in the Serra Gaúcha and who were identified as having HF by the attending physician will be included. Upon discharge, patients will leave the hospital with a date and time to return to the HF Ambulatory. In the first consultation, patients will be invited to participate in the study and will answer a nursing screening instrument and the following instruments: WHOQOL-BREF and ICPT (respectively, quality of life and post-traumatic growth). In order of date and time when signing the informed consent form, patients will be randomized in 1: 1. From the second consultation, the intervention group will be followed up for guidance on the disease and treatment, totaling 12 sessions in 6 months. The control group will go through medical consultations as instructed by the doctor and will not receive intervention for health education by the nurse. After the end of the treatment, the patients will be followed in order to verify the occurrence of new hospitalizations in 6 months and in 1 year. At the end of 1 year the instruments will be replicated. Results: It is expected to enable the patient to remain free of the symptoms of the disease, following the prescribed treatment and being able to recognize any changes that signal an aggravation of the disease. It is hoped that the intervention in health education can decrease the rate of rehospitalization of patients, improve the quality of life and provide greater post-traumatic growth in patients with HF.

DETAILED DESCRIPTION:
Adult patients (≥ or equal to 18 years old), who were admitted to any ward or intensive care unit (ICU) for the cardiology team, and who have been identified as having HF will be included. Octogenarians and / or with communication barriers will be excluded (due to the difficulty of self-management of signs and symptoms, not in line with the objective to be studied) and still not accept to participate in the study. Upon discharge, patients with HF will leave the hospital with a date and time to return to the HF outpatient clinic.

At the time of the first medical consultation, patients will complete a screening instrument (Appendix A) that contains information about: age; sex; breed; origin (city); inpatient for the cardiology team; length of hospital stay; cause of hospitalization; laboratory values (urea and creatinine); echocardiographic data up to 1 year before admission: left ventricular ejection fraction (LVEF); associated comorbidities, medications for continuous use, daily practices related to physical exercise, sodium intake, smoking, body weight, classification according to the New York Heart Association (NYHA), and a brief report on its understanding of the disease (HF) and its strategic control of warning signs and symptoms; After filling in these data, patients will be invited to participate in the study. Those who accept it, signing the IC (Annex B), will answer the following instruments: WHOQOL-BREF and ICPT. In order of date and time when signing the informed consent form, patients will be randomized in 1: 1, with odd numbers designated for treatment A (intervention for self-care) and even numbers designated for treatment B conventional treatment 24.

From the second consultation, patients will be treated differently:

Control Group: The control group will undergo medical consultations as instructed by the attending physician and will not receive intervention for health education by the nurse.

Intervention group:

First, health education will be carried out by the nurse, explaining the importance of daily body weight control, inspecting the ankles for swelling, preventing respiratory diseases (flu vaccine), eating low-salt foods, control of the amount of liquid ingested, the need to follow the schedule and the correct dose of the prescribed drugs. In the third consultation, the patient will be evaluated regarding follow-up with the correct diet, intake of controlled fluids, consistency with the use of medications (explaining the purpose of each). Check with the patient his ability to remain free of the symptoms of the disease, the follow-up of the treatment, if he recognizes any change that signals an aggravation of the disease (explaining about the dangerous signs and symptoms that must be observed by the patient). From the fourth consultation, an explanatory brochure will be delivered which denotes the signs and symptoms that should be observed and when to seek outpatient service in order to avoid an aggravation of the disease by postponing an apparent symptom. Guidance will be given in relation to quality of life, changes in lifestyle, investigating the patient's support network and internal changes in relation to their view of life and spirituality from the diagnosis of the disease.

The consultations will be individual, weekly (Wednesdays), the others, therefore, will be biweekly, extending to the 30/30 days the following, individually in order to observe the difficulties and doubts of each patient. Counting the meetings in a total of 12 in the first 6 months.

After the end of the treatment, the patients will be followed in order to verify the occurrence of new hospitalizations in 6 months and in 1 year. At the end of 12 months, the instruments will be replicated.WHOQOL_BREF: The WHOQOL-BREF consists of 26 questions whose answers follow a Likert scale (from 1 to 5, the higher the score the better the quality of life). Questions 1 and 2 deal with general quality of life. Apart from these two questions (1 and 2), the instrument has 24 more questions which make up 4 domains which are: PHYSICAL, PSYCHOLOGICAL, SOCIAL RELATIONSHIPS and ENVIRONMENT25. (Annex C) Post-Traumatic Growth Inventory (ICPT): Post-traumatic growth consists of the idea that when experiencing an adverse situation, such as becoming ill or worsening health conditions, the person can positively change the way they see and relate with the world. (ICPT) is a self-report scale that evaluates 5 domains, being: Relationship with others (7 items, ex: "I have a clearer idea that I can count on people in times of difficulty"); New possibilities (5 items, ex: "I developed new interests"); Personal Change (4 items, ex: "I know I can handle difficulties better"), Spiritual Change (2 items, ex: "I have a better understanding of spiritual issues") and Greater appreciation of life (3 items, ex: " I get to enjoy each day better "). The responses follow a Likert scale (from 0 to 5, from "I did not experience this change ..." to "I completely experienced this change as a result of the event" 26) (Annex D)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ or equal to 18 years) will be included, who were admitted to any ward or intensive care unit (ICU) of this hospital (for the cardiology team) and who have been identified as having HF indicated by the attending physician via medical records. electronic

Exclusion Criteria:

* Octogenarians and / or communication barriers will be excluded from the analysis (due to the difficulty of self-management of the signs and symptoms, in contrast to the objective to be studied), patients do not accept to participate in the study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Rehospitalisation | 1 year follow up
  record of rehospitalizations due to decompensation in 1 year of follow-up; checked in, yes or no and how many times

SECONDARY OUTCOMES:
WHOQOL BREF | difference between baseline data and at 1 year of follow-up
  It consists of 26 questions whose answers follow a Likert scale (from 1 to 5, the higher the score the better the quality of life), the score therefore varies from 26 to 130 points.
Pos traumatic grown factor | difference between baseline data and at 1 year of follow-up
  It is a series of questions that evaluate the intensity through a likert scale from 0 to 5, the score ranges from 0 to 105.

CONTACTS AND LOCATIONS:
Locations (1):
- Marcia Moura Schmidt, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Oliveira FW, Nunes BP, Lobato FL, Schmidt MM. Psychoeducational Intervention for Reducing Heart Failure Patients' Rehospitalizations and Promoting Their Quality of Life and Posttraumatic Growth at the 1-Year Follow-Up: A Randomized Clinical Trial. Psychosom Med. 2023 Apr 1;85(3):273-279. doi: 10.1097/PSY.0000000000001180. Epub 2023 Feb 26. PMID 36917484